CLINICAL TRIAL: NCT04745559
Title: Optimizing Cellular and Humoral Immunity to Pneumococcus by Vaccination With Pneumococcal 13-valent Conjugate Vaccine Before and After CD19-targeted CAR T-cell Immunotherapy
Brief Title: Optimizing Cellular and Humoral Immunity by Vaccinating With PCV13 Before and After CAR-T Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20571
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large-Cell Lymphoma; Primary Mediastinal Large B-Cell Lymphoma (PMBCL); Transformed Follicular Lymphoma (TFL); High-grade B-cell Lymphoma (HGBCL); Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Pneumococcal Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Pneumococcal conjugate vaccine (PCV13) .5 ml will be administered intramuscularly three times: 7 days (range 4 to 21 days) before apheresis collection and on day +30 (range +21 to +37) and day +90 (range +75 to +115) after CAR T cell infusion.
  Interventions: Biological: Pneumococcal conjugate vaccine (PCV13); Biological: CD19 targeted CAR T Cell Therapy

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine (PCV13) — Licensed heptavalent pneumococcal conjugate vaccine (PCV13, Pneumococcal 13-valent conjugate vaccine
  Other Names: Prevnar 13
Biological: CD19 targeted CAR T Cell Therapy — This is a personalized therapeutic approach that entails removal of T cells from patient's peripheral blood, genetic modification, activation and expansion in vitro to retarget cells against CD19 protein on the surface of B cells, and infusion of the genetically engineered cells back into the patient. CD19 is a surface protein that is expressed on B cells starting from early pre-B cells to mature fully differentiated B cells. Therefore, CD19-targeted CAR T cell therapy can effectively treat refractory B cell lymphomas.

SUMMARY:
The purpose of the study is to evaluate whether receiving the pneumococcal 13-valent conjugate vaccine (PCV13) before and after CD19-targeted CAR T cell therapy will optimize cellular and humoral immunity to pneumococcus.

DETAILED DESCRIPTION:
This is a phase II, single-institution study to investigate if pneumococcal vaccination before and after CD19-targeted CAR T cell therapy elicits cellular and humoral immunity to pneumococcus in patients with relapsed or refractory B cell lymphomas. All the participants will receive the same treatment. Immunoglobulins (IgG) against pneumococcal serotypes not included in the vaccine will be served as an internal control. Treatment includes the same dose (0.5ml) of PCV13 one time prior to apheresis followed by two times after CAR T cell therapy

ELIGIBILITY:
Inclusion Criteria:

* In good health as evidenced by medical history or diagnosed with relapsed or chemotherapy-refractory diffuse large B cell lymphoma (DLBCL), primary mediastinal B cell lymphoma (PMLBCL), transformed follicular lymphoma (TFL) high-grade B cell lymphoma (HGBCL) or Follicular Lymphoma. Patients must be under consideration for treatment with any CD19-targeted CAR T cell therapy, per institutional standards. Patients undergoing active vital organ testing with a planned apheresis date for CAR T cell therapy may be considered eligible.
* Signed informed consent form in accordance with institutional and federal law policies
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, age over 18
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation

Exclusion Criteria:

* Pregnant or lactating woman, as evaluated by serum testing within 2 weeks of administration of the first vaccine. Only women of childbearing potential will undergo serum/urine pregnancy testing. A woman will be considered of childbearing potential unless she is status-post hysterectomy or tubal ligation or without menstrual periods in the preceding 12 months.
* Common variable immunodeficiency or other inherited systemic immunodeficiency syndrome
* History of severe allergy (e.g., anaphylaxis) to any component of pneumococcal conjugate vaccine 7 valent (PCV7), PCV13, or any diphtheria-toxoid containing vaccine.
* Inclusion on a separate trial in which patients may be randomized or otherwise started on maintenance chemotherapies within the first 3 months of CD19-targeted CAR T cell therapy
* Patients with significant psychiatric illness likely to affect compliance, as determined by the treating physician
* Active or uncontrolled infections
* Platelet count <10,000 cells/microliter
* Lymphocyte count <200 cells/microliter
* Intervenous immunoglobulin (IVIG) administration within one month of planned apheresis for collection for CD19-targeted CAR T cell manufacture
* History of PCV13 administration within one month of planned apheresis for collection for CD19-targeted CAR T cell manufacture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Humoral Response Rate -PCV13 vaccine | 90 days post CAR T therapy
  Humoral sero-protection rate elicited by the PCV13 vaccine intervention as measured on day+90 post CART

SECONDARY OUTCOMES:
Increase in PCV13 specific serotype IgG levels | 90 days post CAR T therapy
  PCV13 specific serotype IgG levels on day +90 post CAR T cell therapy as an absolute and as a change from baseline
Increase in On-Specific Serotype IgG levels | 90 days post CAR T therapy
  Non-specific serotype IgG levels on day +90 post CAR T cell therapy as an absolute and as a change from baseline
Response Rate of CD19-targeted CAR T therapy when combined with PCV13 vaccination | 90 days post CAR T therapy
  Percentage of patients whose cancer shrinks or disappears after treatment
Progression Free Survival | at 90 days and 180 days post CAR T therapy
  Progression Free Survival (PFS) from start of treatment to death of any cause, disease progression or relapse of the date of last follow-up, whichever comes first.
Overall Survival | 180 days post CAR T therapy
  Overall Survival (OS):The length of time from the start of treatment until death by any cause

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Locke, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States